CLINICAL TRIAL: NCT06672354
Title: Effects of Non-immersive Virtual Reality Training Compared to Otago Exercise Program on Balance and Spatiotemporal Gait Parameters in Elderly Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/41
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Elderly; Balance; Gait; Virtual Reality
Keywords: Elderly; Balance; Gait; Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Otago Exercise Program Group (Experimental): It includes participants receiving Otago Exercise Program, which consists of stengthening, balance exercises and walking plan.
  Interventions: Procedure: Otago Exercise Program
- Non-Immersive Virtual Reality Group (Experimental): This group involves participants receiving VR training exercises by using Xbox Kinect 360.
  Interventions: Procedure: Non-Immersive Virtual Reality Training

INTERVENTIONS:
Procedure: Otago Exercise Program — 1- Otago Exercise Program: i) This exercise program will consist of strengthening, balance exercises and walking plan. The OEP will be performed according to the following: 5 min warm-up, 10 min resistance training and 15 min balance exercises.
  ii) The strength training protocol targets, on hip abductors, knee flexors, knee extensors, plantarflexors, and dorsiflexors.All exercises will be performed for 10 repetitions. This protocol recommends strength training 3 days per week.
  iii) The balance retraining protocol incorporates various exercises. The exercises progress in difficulty through four levels, with Level 1 being the easiest and Level 4 the most challenging. Balance exercises will progress from holding onto a stable supporting structure such as heavy furniture to perform the exercises independent of the support. The protocol recommends participants to carry out balance exercises 3 days a week.
  iv) Participants will be instructed to walk at their usual pace for 30 minutes, twice
  Arms: Otago Exercise Program Group
Procedure: Non-Immersive Virtual Reality Training — In this interventional group, VR training exercises will be performed by using Xbox Kinect, which includes a Kinect sensor.-The monitor or Tv screen will recognize the movements of participants via camera and infra-red motion sensors.-In order to perform simulated exercises in each session, the participant will be positioned at 1.5-2 meter from the monitor or TV screen.-The virtual reality training exercises will include Kinect Adventure games (Rally Ball, 20,000 leaks, Reflex Ridge) and Sports pack 1 games (Super Saver, Target Kick, Body ball).-Exercises will be continued for 30-45 minutes each session, for 3 alternate days per week for a total period of 12 weeks.
  Arms: Non-Immersive Virtual Reality Group

SUMMARY:
Falling is a serious concern for the growing elderly population due to age-related decline in physical function, leading to injuries, loss of independence, and a decline in overall well-being.

The Otago Exercise Program (OEP), for the elderly consists of lower limb strengthening and balance exercises, leading to better strength, balance, and reduced fear of falling.

The interactive and game-like nature of VR training can make it more engaging and motivating for older adults. It can provide challenging and engaging approach to exercise that can help to improve stability, enhance quality of life and reduce the risk of fall.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the effects of Non-Immersive VR training and Otago exercise program on spatiotemporal gait parameters in elderly population.
2. To determine the effects of Non-Immersive VR training and Otago exercise program on balance in elderly population.
3. To determine the effects of Non-Immersive VR training and Otago exercise program on lower limb strength of elderly population.
4. To determine the effects of Non-Immersive VR training and Otago exercise program on fear of fall in elderly population.

HYPOTHESIS:

Alternate Hypothesis:

1. There is statistically significant difference between non-immersive virtual reality training and Otago exercise program on spatiotemporal gait parameters in elderly population.
2. There is statistically significant difference between non-immersive virtual reality training and Otago exercise on balance in elderly population.
3. There is statistically significant difference between non-immersive virtual reality training and Otago exercise on lower limb strength in elderly population.
4. There is statistically significant difference between non-immersive virtual reality training and Otago exercise on fear of fall in elderly population.

Null Hypothesis:

1. There is no statistically significant difference between non-immersive virtual reality training and Otago exercise program on spatiotemporal gait parameters in elderly population.
2. There is no statistically significant difference between non-immersive virtual reality training and Otago exercise on balance in elderly population.
3. There is no statistically significant difference between non-immersive virtual reality training and Otago exercise on lower limb strength in elderly population.
4. There is no statistically significant difference between non-immersive virtual reality training and Otago exercise on fear of fall in elderly population.

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Multidisciplinary Lab in FUCP. Study duration: 1 year

Selection Criteria:

Inclusion Criteria

1. Age 55 years and above
2. Male and female both
3. Able to independently ambulate, without the assistance of a walking aid.
4. Participants that are able to maintain upright position with eyes open and eyes close for 10 seconds in standing position

Exclusion Criteria

1. Wheel-chair bound elderly
2. Diagnosed with neurological disorder
3. Severe cognitive impairment (MMSE scoring of 17 or <17)
4. Recent orthopedic trauma
5. Severe degenerative conditions

Technique: Non probability Purposive Sampling

Outcome Measures:

Data will be collected on Demographics and general information. Data will be collected using Mini-BESTEST scale, 10 Meter walk test, 30 sec sit to stand test, The Fall Efficacy Scale International

Expermental Group (A) =This group will recive Otago Exercise Program training outcomes will be measured at baseline, on 4th, 8th and at 12th week of treatment.

Data analysis techniques:

Experimental Group (B) = This group will receive Non-Immersive Virtual Reality training using Xbox Kinect 360. Their outcomes will be measured at baseline, on 4th, 8th and at 12th week of treatment.

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study within the community.

A printed questionnaire will be provided to the patients after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

While the Otago Exercise Program (OEP) has established itself as a highly effective intervention for improving balance and reducing fall risk in older adults, the emergence of non-immersive Virtual Reality (VR) training introduces a potentially complementary approach.

However, despite both offering multi-component interventions targeting fall risk factors, a lack of conclusive evidence exists regarding their differential impact on balance and gait parameters.

Our study addresses this critical gap in the literature by directly comparing the efficacy of non-immersive VR training against the OEP.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years and above
* Male and female both
* Able to independently ambulate, without the assistance of a walking aid.
* Participants that are able to maintain upright position with eyes open and eyes close for 10 seconds in standing position

Exclusion Criteria:

* Wheel-chair bound elderly
* Diagnosed with neurological disorder
* Severe cognitive impairment (MMSE scoring of 17 or <17)
* Recent orthopedic trauma
* Severe degenerative conditions

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Balance | 12 weeks
  The Mini-BESTest includes 14 items that examine performance tasks related to dynamic balance. The test has a maximum score of 28 points from 14 items that are each scored from 0-2.
Gait Speed | 12 weeks
  he 10 Meter Walk Test, will be used to assess walking speed in meters per second over a short distance. Using the data from the test i.e. time taken to complete distance and step count, gait speed will be evaluated based on the given formula: Distance walked/time(sec)
Cycle Time | 12 weeks
  The 10 Meter Walk Test, will be used to assess walking speed in meters per second over a short distance. Using the data from the test i.e. time taken to complete distance and step count, cycle time will be evaluated based on the given formula: Time(sec) x 2 /No. of steps
Stride Length | 12 weeks
  The 10 Meter Walk Test, a performance measure will be used to assess walking speed in meters per second over a short distance. Using the data from the test i.e. time taken to complete distance and step count, stride length will be evaluated based on the given formula: gait speed (m/s) x cycle time(sec)
Cadence | 12 weeks
  The 10 Meter Walk Test, a performance measure will be used to assess walking speed in meters per second over a short distance. Using the data from the test i.e. time taken to complete distance and step count, cadence will be evaluated based on the given formula: No of steps x 60/time(sec)
Leg Strength | 12 weeks
  The 30 Second Sit to Stand Test will be used to test leg strength and endurance in older adults. The test stand involves recording the number of stands a person can complete in 30 seconds.
Fear of Fall | 12 weeks
  The Falls Efficacy Scale International, measure of "fear of falling" or "concerns about falling. It is a 16-item questionnaire, the item scores are summed up to obtain a total, with a score ranging from minimum 16 to maximum 64.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan